CLINICAL TRIAL: NCT02781350
Title: To Study the Effect of High Fat High Carbohydrate Meal on Oxidative Load, Inflammatory Mediators and Insulin Resistance in Normal and Obese Subjects
Brief Title: Anti-inflammatory Effects of Fiber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Paresh Dandona, SUNY Distinguished Professor, University at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1955
Record Dates: First submitted 2016-04-25; First posted 2016-05-24 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Postprandial Inflammation
Keywords: high fat diet; insulinogenesis; Fiber; inflammation
MeSH Terms: conditions — Inflammation | interventions — Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fat high carbohydrate (HFHC) meal (Placebo Comparator): Subjects will consume a HFHC meal. HFHC meal includes egg muffin and sausage muffin sandwiches and two hash browns which contain 88g carbohydrates, 51 g fat (33% saturated) and 34 g protein (carbohydrates 41%, protein 17%, and fat 42%). 35 ml of blood will be obtained at 1h ,2h,3h and 4 h and 5 ml at 15 min,30 min,45 min,75 min and 90 min . A total of 165 ml (11 tablespoon) blood will be collected.
  Interventions: Other: HFHC meal
- HFHC meal plus Fiber (Experimental): HFHC meal includes egg muffin and sausage muffin sandwiches and two hash browns which contain 88g carbohydrates, 51 g fat (33% saturated) and 34 g protein (carbohydrates 41%, protein 17%, and fat 42%). Subjects will also receive FiberOne Original cereal 14 grams (half cup) before and after the HFHC meal. 35 ml of blood will be obtained at 1h ,2h,3h and 4 h and 5 ml at 15 min,30 min,45 min,75 min and 90 min . A total of 165 ml (11 tablespoon) blood will be collected.
  Interventions: Dietary Supplement: HFHC MEAL plus Fiber

INTERVENTIONS:
Other: HFHC meal — 900 Cal high fat high carbohydrate fast food meal (HFHC). meal includes egg muffin and sausage muffin sandwiches and two hash browns which contain 88g carbohydrates, 51 g fat (33% saturated) and 34 g protein (carbohydrates 41%, protein 17%, and fat 42%).
  Arms: High fat high carbohydrate (HFHC) meal
Dietary Supplement: HFHC MEAL plus Fiber — 900 Cal high fat high carbohydrate fast food meal containing egg muffin and sausage muffin sandwiches and two hash browns which contain 88g carbohydrates, 51 g fat (33% saturated) and 34 g protein (carbohydrates 41%, protein 17%, and fat 42%).with FiberOne Original cereal 14 grams (half cup) each before and after the HFHC meal
  Arms: HFHC meal plus Fiber

SUMMARY:
The main objective of this research is to investigate the effect of addition of fiber on the high fat high carbohydrate (HFHC) meal induced inflammation and oxidative stress mechanisms at the molecular level in humans, in vivo. The investigators have previously shown that the intake of one HFHC meal leads to an increase in oxidative stress and inflammation. HFHC meal also induces an increase in the expression of suppressor of cytokine signaling- 3 (SOCS-3) in the mononuclear cells (MNC), which interferes with insulin signal transduction and contributes to the pathogenesis of insulin resistance. In contrast, an American heart association (AHA) meal rich in fruits and fiber does not induce these effects. These observations are important since HFHC meal not only induces oxidative stress and inflammation but also lays the foundations of a potentially greater insulin resistance through the induction of SOCS-3, TLR-4 and TLR-2.

DETAILED DESCRIPTION:
The main objective of this research is to investigate the effect of high fat high carbohydrate (HFHC) meal on inflammatory mechanisms at the molecular level in humans, in vivo versus HFHC meal plus fiber. HFHC meal includes egg muffin, sausage muffin sandwiches and two hash browns. The Investigators have previously shown that the intake of one HFHC meal leads to an increase in reactive oxygen species (ROS) generation and the expression of p47, the key subunit of NADPH oxidase, with a concomitant increase in intranuclear nuclear factor κB (NFkB) binding. More recently, the investigators have also shown that HFHC meal leads to an increase in plasma endotoxin (lipopolysaccharide, LPS) concentrations along with an increase in the expression of Toll like receptor-4 (TLR-4), the receptor for endotoxin, and TLR-2, the receptor for several products of Gram positive bacteria. In addition, it also causes an increase in lipopolysaccharide binding protein (LBP), the protein which facilitates the binding of LPS to CD14 and TLR-4. Finally, HFHC meal also induces an increase in the expression of suppressor of cytokine signaling- 3 (SOCS-3) in the mononuclear cells (MNC) (1), which interferes with insulin signal transduction and contributes to the pathogenesis of insulin resistance. In contrast, an AHA meal does not induce these effects. These observations are important since HFHC meal not only induces oxidative stress and inflammation but also lays the foundations of (2) a potentially greater response to an inflammatory challenge through the induction of an increase in LPS concentrations and the expression of TLR-4 and TLR-2; and (3) insulin resistance through the induction of SOCS-3, TLR-4 and TLR-2.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 80 years of age
* Subject will be available for duration of the study and willing to comply with all study requirements
* Written and informed consent signed and dated
* Nonsmoker

Exclusion Criteria:

* Coronary artery disease (CAD): documented by history of myocardial infarction, angioplasty/stent placement, angina, exercise EKG positive for ischemia or angiographic evidence of CAD
* Patient on non-steroidal anti-inflammatory drugs or steroids
* Hepatic disease (transaminase > 3 times normal)
* Renal impairment (serum creatinine > 1.5 mg/dl)
* History of drug or alcohol abuse
* Participation in any other concurrent clinical trials
* Use of an investigational agent or therapeutic regimen within 30 days of study
* Pregnancy
* Premenopausal women who are trying to be pregnant
* Anemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
effect of addition of fiber on the relative change of NF-Kappa B | Baseline and 1 week
  The investigators hypothesize that addition of fiber intake will suppress NF-kappa B after HFHC meal. Therefore, changes in NF-kappa B activity will be compared as percent change form baseline after HFHC meal with or without fiber in lean and obese subjects

SECONDARY OUTCOMES:
effect of addition of fiber on Changes in ROS generation. | Baseline and 1 week
  Changes in Reactive oxygen species (ROS) generation between the 2 visits (HFHC meal with or without fiber) will be compared as percent change from baseline.
effect of addition of fiber on Changes in TLR-4 mRNA expression in MNC | Baseline and 1 week
  Changes in TLR-4 mRNA expression in MNC between the 2 visits (HFHC meal with or without fiber) will be compared as percent change from baseline.
effect of addition of fiber on Changes in SOCS-3 mRNA expression in MNC | Baseline and 1 week
  Changes in SOCS-3 mRNA expression in MNC between the 2 visits (HFHC meal with or without fiber) will be compared as percent change from baseline.
effect of addition of fiber on Changes in insulin secretion between the 2 visits (HFHC meal with or without fiber) will be compared as percent change from baseline. | Baseline and 1 week
  Changes in insulin concentrations between the 2 visits (HFHC meal with or without fiber) will be compared as percent change from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- ECMC Ambulatory Center, 3rd Floor, Buffalo, New York, United States